CLINICAL TRIAL: NCT00284583
Title: Comparison of Corticosteroid and Ethanol Injection Therapy in the Treatment of Morton's Neuroma
Brief Title: Comparison of Alcohol and Steroid Injection for Treating Morton's Neuroma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brown University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0061-05
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2006-01

CONDITIONS: Morton's Neuroma
Keywords: Morton's Neuroma; Alcohol; Steroid
MeSH Terms: conditions — Morton Neuroma | interventions — Ethanol

INTERVENTIONS:
Drug: Injection of Steroid into Foot
Drug: Injection of Alcohol into Foot
Drug: Injection of Lidocaine into Foot

SUMMARY:
Interdigital neuroma is a painful forefoot disorder characterized by plantar pain and toe paresthesias thought to result from entrapment of the interdigital nerve by the overlying transverse metatarsal ligament. Multiple treatments have been recommended for this condition and range from modification of shoe wear to surgical excision of the painful nerve. Serial ethanol injection therapy has been reported to be an effective alternative to surgical excision. However, despite wide adoption of this treatment, no randomized, double blinded, placebo-controlled study exists to verify the efficacy of this treatment in comparison to longer standing similar therapies, such as corticosteroid injection.

120 patients from one Orthopaedic group's foot and ankle offices with single foot neuromas and no previous history of neuroma or foot disorder treatment will be selected for the study. These patients will be randomized to three treatments, specifically lidocaine injection, corticosteroid injection, or ethanol injection. Outcomes will be assessed at 3, 6 and 12 month time points using validated questionnaires as well as a non-validated disease specific questionnaire. Primary endpoint will be graded change in the physical function portion of the SF-36 form. Secondary endpoints will be the graded change in the McGill Short Form for Pain and ultimate satisfaction with treatment as assessed by a non-validated questionnaire designed for Morton's neuroma symptoms.

DETAILED DESCRIPTION:
Interdigital neuroma, or Morton's Neuroma, is a painful forefoot disorder characterized by plantar pain and paresthesias radiating to toes. The condition was first described in 1845 by Lewis Durlacher as a painful "neuralgic affection" of the plantar nerve between the third and fourth metatarsals. T.G. Morton, in 1876, attributed the painful symptom complex to a "neuroma." His observation was confirmed by Hoadley who, in 1893, performed a curative excision of a "neuroma" between the third and fourth metatarsals.

Current understanding of interdigital neuroma is based on Gauthier's conclusion in 1979 that the symptom complex was a result of an entrapment neuropathy of the interdigital nerve by the overlying transverse metatarsal ligament. Presently, no definitive single etiology has been confirmed. Additional potential pathoetiologies include the aberrant anatomy of the plantar nerve in this location, trauma and extrinsic mass effect above or below the level of the transverse metatarsal ligament.(3,6) The histological appearance of the affected nerve, however, is consistent and suggests that "neuroma" is a misnomer for this condition. The nerve tissue demonstrates demyelination and deposition of amorphous eosinophilic material, but no exuberant proliferation of nerve endings characteristic of neuroma.(3)

Multiple treatments have been recommended for the management of interdigital neuroma. The usual algorithm begins with an attempt at conservative therapy consisting of shoe wear modifications and the application of a metatarsal pad. Failure of conservative management may prompt a trial of corticosteroid injections.(8) Persistent symptoms ultimately require surgical excision or division of the transverse metatarsal ligament, both of which have good long term outcomes in literature.(2,7)

Recently, serial ethanol injection therapy has been reported to be an effective alternative to surgical excision and has been widely adopted in the treatment of Morton's neuroma. Dockery et. al. reported 89% success rate in a series of 100 consecutive patients treated with 3 to 7 injections of 4% ethanol solutions with an average follow-up of 13 months. Fanucci and Masala reported a 90% success rate at 10 month follow-up after 3 to 7 injections of 30% alcohol in a consecutive series of 40 patients. However, none of these studies were performed in a randomized, double blinded fashion with adequate controls. Therefore, no scientifically valid conclusions concerning treatment efficacy can be made.

The proposed study investigates alcohol sclerosing therapy for the treatment of Morton's neuroma in a randomized, double-blinded, placebo-controlled clinical trial. The primary end point will be evaluation of patient physical function according to the standardized SF-36 questionnaire after the treatment period. Secondary end points include evaluation of pain and satisfaction levels after treatment using, respectively, a standardized and a novel questionnaire.

ELIGIBILITY:
Inclusion Criteria:

2 months of 2 or more of the following

* Plantar pain increased by walking localized to the 2nd and 3rd interspaces
* Relief of pain by resting
* Pain radiating into toes
* Numbness in toes or foot
* Cramping in toes and foot

  2 or More of the Following physical Findings
* Plantar tenderness
* Radiation of elicited pain into the toes
* Palpable plantar mass
* Numbness in toes
* Exacerbation of symptoms with Mulder's maneuver

Exclusion Criteria:

* Past treatment for Morton's neuroma or had prior foot surgery.
* Concurrent conditions such as hallux valgus, metatarsalgia, lesser toe abnormalities, atraumatic synovitis of metatarsophalangeal joint and other foot and ankle based nerve compression neuropathies.
* Further, patients with neuroma symptoms in the 1st and 4th interspaces.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-05

PRIMARY OUTCOMES:
1. Pain Scale
2. Physical function scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Digiovanni, MD, Principal Investigator — Rhode Island Hospital, Brown Medical School
Locations (1):
- Rhode Island Hospital Orthopaedic Clinic, Providence, Rhode Island, United States

REFERENCES:
- [Background] Bennett GL, Graham CE, Mauldin DM. Morton's interdigital neuroma: a comprehensive treatment protocol. Foot Ankle Int. 1995 Dec;16(12):760-3. doi: 10.1177/107110079501601204. PMID 8749346
- [Background] Bradley N, Miller WA, Evans JP. Plantar neuroma: analysis of results following surgical excision in 145 patients. South Med J. 1976 Jul;69(7):853-4. PMID 941051
- [Background] Dockery GL. The treatment of intermetatarsal neuromas with 4% alcohol sclerosing injections. J Foot Ankle Surg. 1999 Nov-Dec;38(6):403-8. doi: 10.1016/s1067-2516(99)80040-4. PMID 10614611
- [Background] Fanucci E, Masala S, Fabiano S, Perugia D, Squillaci E, Varrucciu V, Simonetti G. Treatment of intermetatarsal Morton's neuroma with alcohol injection under US guide: 10-month follow-up. Eur Radiol. 2004 Mar;14(3):514-8. doi: 10.1007/s00330-003-2057-7. Epub 2003 Oct 3. PMID 14531002